CLINICAL TRIAL: NCT01985061
Title: Prospective and Multicentre Evaluation of 3 Different Doses of IV Busulfan Associated With Fludarabine and Thymoglobuline in the Conditioning of Allogeneic Stem Cell Transplantation (SCT) From a Matched Related or Unrelated Donor in Patients With Poor Prognosis Myeloid Malignancies
Brief Title: Evaluation of 3 Different Doses of IV Busulfan
Acronym: AAA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAA-IPC2011-003
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: Myelodysplasic syndrome; Acute Myeloid leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BX2 (Active Comparator): Fludarabine (Fludara®): 30 mg/m2 on D-6, D-5, D-4, D-3 and D-2 Busulfan IV (Busilvex®) : 3.2 mg/kg/d on D-4 and D-3 Thymoglobuline®: 2.5 mg/kg/d on D-3 and D-2
  Interventions: Drug: BX2
- BX3 (Experimental): Fludarabine (Fludara®): 30 mg/m² on D-6, D-5, D-4, D-3 and D-2 Busulfan IV (Busilvex®) : 3.2 mg/kg/d on D-5, D-4 and D-3 Thymoglobuline® : 2.5 mg/kg/d on D-3 and D-2
  Interventions: Drug: BX3
- BX4-Suspended (Active Comparator): Fludarabine (Fludara®): 30 mg/m²on D-6, D-5, D-4, D-3 and D-2 Busulfan IV (Busilvex®) : 3.2 mg/kg/d on D-6, D-5, D-4 and D-3 Thymoglobuline® : 2.5 mg/kg/d on D-3 and D-2
  Interventions: Drug: BX4-Suspended

INTERVENTIONS:
Drug: BX2
  Other Names: Busulfan Intravenous 2 days at 3.2 mg/kg/d
  Arms: BX2
Drug: BX3
  Other Names: Busulfan Intravenous 3 days
  Arms: BX3
Drug: BX4-Suspended — Suspended
  Other Names: Busulfan intravenous 4 days
  Arms: BX4-Suspended

SUMMARY:
Albeit the safety of the stem cell transplantation procedure has been greatly improved, further refining the intensity of the conditioning is an important issue to explore, especially in patients with poor prognosis, the goal being to maintain the very favorable safety profile and improve the disease control. This is the goal our prospective trial; we aim to prospectively evaluate in a prospective multicenter trial the efficacy of different conditioning regimens in patients with high-risk myeloid malignancies.

The study is a phase II trial randomizing patients between a prospective active control arm (BX2) and two experimental arms (BX3 and BX4). A standard group was kept in this clinical trial in order to avoid the limitations induced by the comparison with historical controls in the context of continuously improving practice. Each experimental arm will be conducted in parallel according to a standard phase II trial design.

In addition, this trial will associate four ancillary studies to the main clinical objective: 1/ a prospective assessment of the quality of life of the patients over a period of 2 years 2/ an analysis of the cost effectiveness of the procedure, assessed over a period of 2 years 3/ an observational busulfan pharmacokinetic study 4/ a busulfan pharmacogenomic study

ELIGIBILITY:
Inclusion Criteria:

1. Patients with poor prognosis myeloid malignancies:

   * Myelodysplastic syndrome,
   * Acute Myeloid Leukemia (AML) beyond Complete Response (CR1),
   * CR1 AML with poor risk cytogenetics
2. Adult patients: aged ≥ 55 years up to 65 or < 55 years not eligible for myeloablative conditioning regimen based on Total Body Irradiation (TBI) or double alkylating agent combinations.
3. Availability of a HLA identical sibling or matched unrelated donor (10/10)
4. Affiliation to social security
5. Written Informed Consent

Exclusion Criteria:

1. History of previous Allo-Hematological Stem Cell Transplantation (HSCT)
2. HIV positivity
3. Signs of chronic active hepatitis B and/or C
4. Evolutive psychiatric disease
5. Concomitant neoplastic disease
6. Pregnant or lactating woman or without contraception (for child bearing potential wom-en)
7. Usual contra-indications for Allo-HSCT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2026-07-07 (Estimated); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
Time to progression or death | up to 2 years
  2-year progression free survival rates

SECONDARY OUTCOMES:
Time to neutrophil>0.5G/l and platelets>50G/l | up to 2 months
  hematologic recovery
Graft versus host disease | up to 2 years
relapse | up to 2 years
Occurrence of grade 3-4 adverse events according the CTC-AE v4.0 scale | up to 6 months
  safety

CONTACTS AND LOCATIONS:
Overall Officials: Didier BLAISE, MD PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France

REFERENCES:
- [Derived] Wanquet A, Crocchiolo R, Furst S, Granata A, Faucher C, Devillier R, Harbi S, Lemarie C, Calmels B, Vey N, Weiller PJ, Chabannon C, Castagna L, Blaise D, El-Cheikh J. The efficacy and safety of a new reduced-toxicity conditioning with 4 days of once-daily 100 mg/m(2) intravenous busulfan associated with fludarabine and antithymocyte globulins prior to allogeneic stem cell transplantation in patients with high-risk myelodysplastic syndrome or acute leukemia. Leuk Lymphoma. 2016 Oct;57(10):2315-20. doi: 10.3109/10428194.2016.1146948. Epub 2016 Feb 17. PMID 26885686
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr